CLINICAL TRIAL: NCT02582749
Title: Androgen Deprivation Therapy With or Without Radium-223 Dichloride in Patients With Newly Diagnosed Metastatic Prostate Cancer With Bone Metastases: Hoosier Cancer Research Network GU13-170
Brief Title: Androgen Deprivation Therapy +/- Radium-223 Dichloride in Metastatic Prostate Cancer With Bone Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding withdrawn
Sponsor: Ajjai Alva, MD (Other)
Collaborators: Hoosier Cancer Research Network (Other); Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry)
Responsible Party: Sponsor-Investigator, Ajjai Alva, MD, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GU13-170
Record Dates: First submitted 2015-10-16; First posted 2015-10-21 (Estimated); Results first posted 2019-07-09 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Prostate Cancer; Bone Metastases; Prostate Neoplasms
Keywords: Androgen Deprivation Therapy; Androgen Receptor Antagonist; Radium-223 Dichloride; Placebo
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Gonadotropin-Releasing Hormone; bicalutamide; radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Arm A (Active Comparator): All subjects will receive LHRH agonist/antagonist per dosage and route of administration specified by the treating physician. Bicalutamide, 50mg, PO will be administered daily. Cycles will be 28 days.
  Interventions: Drug: LHRH agonist/antagonist; Drug: Bicalutamide
- Experimental Arm B (Experimental): All subjects will receive LHRH agonist/antagonist per dosage and route of administration specified by the treating physician. Bicalutamide, 50mg, PO will be administered daily. Cycles will be 28 days. Radium-223 dichloride, 50 kBq/kg body weight, will be administered as a bolus intravenous (IV) injection at intervals of every 28 days for up to 6 cycles.
  Interventions: Drug: LHRH agonist/antagonist; Drug: Bicalutamide; Radiation: Radium-223 dichloride

INTERVENTIONS:
Drug: LHRH agonist/antagonist — Treating physician will determine LHRH agonist/antagonist, dosage and route of administration, per package insert, during each 28-day cycle.
  Other Names: Per treating physician
Drug: Bicalutamide — Bicalutamide, 50 mg Oral (PO) will be administered daily in each 28-day cycle.
  Other Names: Casodex
Radiation: Radium-223 dichloride — Radium-223 dichloride, 50 kBq (1.35 microcurie) per kg body weight intravenous (IV bolus) every 28 days for 6 injections
  Arms: Experimental Arm B

SUMMARY:
Newly diagnosed metastatic prostate cancer subjects with bone metastases will be accrued to this stratified randomized 2-arm Phase II trial. Subjects will be randomized 1:2 to ADT or ADT with Radium-223 dichloride respectively.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center, randomized trial.

STRATIFICATION FACTORS:

Subjects will be stratified based on serum total alkaline phosphatase at baseline and extent of disease (described below). Randomization will occur within stratification group.

* Extent of Disease: <6 skeletal metastases with no visceral metastases versus ≥6 skeletal metastases or visceral metastases.
* Serum total alkaline phosphatase at baseline: normal vs abnormal. Abnormal alkaline phosphatase is defined as > 130 IU/L.

Early Induction or Late Induction status will not be a stratification criterion.

TREATMENT SCHEDULE: CONTROL ARM A

All subjects will receive androgen deprivation therapy with a LHRH agonist (any LHRH agonist such as leuprolide acetate or goserelin acetate is acceptable) or a LHRH antagonist (degarelix) or bilateral orchiectomy, with dosage determined by the treating physician. Route of administration and cycle days will be administered as per package insert. Androgen deprivation therapy with LHRH agonist or LHRH antagonist will be given continuously.

All subjects will receive bicalutamide, 50 mg Oral (PO) Daily

TREATMENT SCHEDULE: EXPERIMENTAL ARM B

All subjects will receive androgen deprivation therapy with a LHRH agonist (any LHRH agonist such as leuprolide acetate or goserelin acetate is acceptable) or a LHRH antagonist (degarelix) or bilateral orchiectomy, with dosage determined by the treating physician. Route of administration and cycle days will be administered as per package insert. Androgen deprivation therapy with LHRH agonist or LHRH antagonist will be given continuously.

All subjects will receive bicalutamide, 50 mg oral (PO) daily

All subjects will receive Radium-223 dichloride, 50 kBq (1.35 microcurie) per kg body weight, intravenous (IV bolus) every 28 days for 6 injections

The following laboratory values must be obtained within 28 days prior to registration for protocol therapy:

Hematopoietic:

* Hemoglobin (Hgb) ≥ 8.0 g/dL (80 g/L) without packed RBC transfusion
* Platelets ≥ 100 K/mm3
* Absolute neutrophil count (ANC) ≥ 1.5 K/mm3

Hepatic:

* Total Bilirubin ≤ 2 x institutional upper limit of normal (ULN) except subjects with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL
* Aspartate aminotransferase (AST, SGOT) ≤ 2.5 x institutional ULN (≤ 5 x institutional ULN in the presence of liver metastases).
* Alanine aminotransferase (ALT, SGPT) ≤ 2.5 x institutional ULN (≤ 5 × institutional ULN in the presence of liver metastases).

Renal:

* Estimated Creatinine Clearance by Cockcroft-Gault formula ≥ 30 mL/min

ELIGIBILITY:
Inclusion Criteria:

* All subjects or their legally authorized representative must be informed of the investigational nature of the study and provide written informed consent and HIPAA authorization for release of personal health information before performance of any study related procedure not part of routine medical care. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Men ≥ 18 years of age at the time of informed consent.
* Histological or cytological evidence of prostate adenocarcinoma.
* All subjects must have radiologic or pathologic evidence of ≥ 2 skeletal lesions with or without pain at baseline on bone scan or axial imaging or 1 skeletal lesion and bone pain within 28 days prior to the registration.
* All subjects must have a radiographic assessment (chest or abdominal/pelvic CT or MRI) within 28 days prior to registration but do not need to have measurable disease.
* ECOG (Eastern Cooperative Oncology Group) Performance Status of 0-2 within 28 days prior to registration. ECOG Performance Status of 3 will only be allowed if judged by the treating investigator as attributable exclusively to bone pain.
* Subjects must fall into one of the two populations below:
* EARLY INDUCTION GROUP: Subjects who have started androgen deprivation therapy (luteinizing hormone-releasing hormone (LHRH) agonist or antagonist therapy with or without an anti-androgen agent) a maximum of 28 days before registration and who otherwise meet all the eligibility criteria.
* LATE INDUCTION GROUP: Subjects who have NOT started any androgen deprivation therapy (luteinizing hormone-releasing hormone (LHRH) agonist or antagonist therapy with or without an antiandrogen agent).
* Anti-androgen receptor antagonist therapy must be bicalutamide. Subjects already started on other anti-androgens must be willing to switch over to bicalutamide.
* Any prior androgen-deprivation therapy or finasteride as neoadjuvant or adjuvant therapy or for biochemical recurrence must have been discontinued at least 6 months prior to registration.
* Prior surgical treatment for prostate cancer is allowed but must have been completed at least 14 days prior to registration and any toxicity from such therapy must have recovered to ≤ grade 1 per CTCAE version 4 criteria by the time of registration.
* All subjects, including those who are surgically sterilized, must be willing to use an effective method of contraception (barrier method of birth control or abstinence) from the time informed consent is signed until 6 months after completion of protocol therapy.
* Subjects must consent to bank whole blood, serum, plasma for future unspecified studies.

Exclusion Criteria:

* Prior cytotoxic chemotherapy for metastatic prostate cancer. Prior cytotoxic chemotherapy with curative intent in the neoadjuvant or adjuvant setting is allowed but must have been completed at least 6 months prior to registration. No cytotoxic chemotherapy is allowed during protocol specified therapy.
* Prior concomitant therapy with ketoconazole, aminoglutethimide or abiraterone acetate or enzalutamide (MDV3100) or intent to treat with the above. Concurrent megestrol for hot flashes is allowed.
* Prior or ongoing bisphosphonate (e.g,. zoledronic acid) or RANKL inhibitor (e.g. denosumab) use is NOT allowed except when used solely for osteoporosis and strictly per guidelines for that indication. Bisphosphonate or RANKL inhibitor cannot be initiated for any indication during protocol specified therapy without consent of the sponsor-investigator of the study.
* Prior systemic radiotherapy with strontium-89, samarium-153, rhenium-186 or rhenium-188.
* Diagnosis of aplastic anemia, pure red cell aplasia, myelodysplasia or any of the other bone marrow failure states.
* Any neuroendocrine differentiation including small cell carcinoma on histology or cytology.
* No prior malignancy except for non-melanomatous skin cancer or non-muscle invasive bladder cancer or adequately treated Stage I or II cancer (adequacy at discretion of treating investigator) from which the subject is currently in complete remission, or any other cancer from which the subject has been disease-free for at least 3 years.
* History of or active CNS metastasis (brain, leptomeningeal or cord compression). Brain imaging studies are not required for eligibility if the subject has no neurologic signs or symptoms suggestive of brain metastasis. Subjects with neurological symptoms are recommended to undergo a head CT scan (with or without intravenous contrast) or brain MRI (with or without intravenous contrast) to exclude brain metastasis. If brain imaging studies are performed, they must be negative for CNS disease. Skull bone involvement without neurological impact by prostate cancer is allowed.
* Treatment with any other investigational agent within 28 days prior to registration. Subjects must not be treated with any other investigational agent while on protocol specified therapy.
* Prior hemibody external radiation. Any external radiation therapy must have been completed at least 14 days prior to registration. Any toxicity from such therapy must have recovered to ≤ grade 1 per CTCAE version 4 criteria by the time of registration.
* Clinically significant infections as judged by the treating investigator. Subjects must not have been diagnosed with human immunodeficiency virus (HIV) infection, active chronic hepatitis B or C, life-threatening illness unrelated to cancer, or any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with participation in this study. Subjects should be tested for hepatitis B or C or HIV infection during screening only if they are considered by the investigator to be at high risk for these infections.
* Known hypersensitivity to bicalutamide.
* Known gastrointestinal (GI) disease or procedure that could interfere with the GI absorption or tolerance of bicalutamide, including difficulty swallowing oral medications.
* Grade III/IV cardiac disease as defined by the New York Heart Association Criteria (i.e., subjects with cardiac disease resulting in marked limitation of physical activity or resulting in inability to carry on any physical activity without discomfort), symptomatic pulmonary embolism within 3 months, unstable angina pectoris, myocardial infarction within 6 months, or serious uncontrolled cardiac arrhythmia as determined by the treating physician.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2017-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajjai Alva, M.D., Study Chair — Hoosier Cancer Research Network
Locations (12):
- United States (12):
  - University of Arizona Cancer Center at Dignity Health St. Joseph's, Phoenix, Arizona
  - Illinois CancerCare, P. C., Peoria, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers, Indianapolis, Indiana
  - University of Iowa Hopital and Clinics, Iowa City, Iowa
  - University of Michigan Health System, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Metro Health Cancer Center, Wyoming, Michigan
  - GU Research Network, LLC, Omaha, Nebraska
  - Integrated Medical Professionals, PLLC, Lake Success, New York
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Clement J. Zablocki VA Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Arm A | Experimental Arm B
Started | 5 | 11
Completed | 0 | 0
Not Completed | 5 | 11
Not completed — Study terminated by funder | 5 | 10
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm A | Experimental Arm B | Total
Number analyzed (Participants) | 5 | 11 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 2 | 7 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 11 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 11 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 11 | 16
Extent of Disease [Count of Participants; unit: Participants]
  <6 skel met, no visc met, total alk phos<=130 IU/L | 2 | 5 | 7
  <6 skel met, no visc met, total alk phos >130IU/L | 1 | 1 | 2
  >=6 skel met or visc met, total alk phos <=130IU/L | 1 | 4 | 5
  >=6 skel met or visc met, total alk phos >130IU/L | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Radiological Progression-Free Survival (rPFS)
Description: rPFS assessed using Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1) to compare outcomes of subjects on experimental arm vs control arm
Time Frame: From date of randomization to disease progression or death from any cause, up to a maximum of 24 months.
Population: Data was not collected or analyzed for this objective due to the termination of the study by the funder
Arm/Group | Control Arm A | Experimental Arm B
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug, Graded According to NCI Common Terminology Criteria for Adverse Events v 4.0 (CTCAE)
Description: The intensity of AEs for subjects on both arms graded according to CTCAE v4.0 on a five-point scale (Grade 1 to 5: Mild, Moderate, Severe, Life-threatening and Death)
Time Frame: From date of first dose until 30 days after the last treatment, assessed for a maximum of 24 months
Population: Data was not collected or analyzed for this objective due to the termination of the study by the funder
Arm/Group | Control Arm A | Experimental Arm B
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to First Skeletal-Related Event (SRE)
Description: SRE of subjects on both arms assessed by bone scan or axial imaging
Time Frame: From date of first dose until 30 days after the last treatment, assessed for a maximum of 24 months
Population: Data was not collected or analyzed for this objective due to the termination of the study by the funder
Arm/Group | Control Arm A | Experimental Arm B
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Secondary Neoplasms
Description: Secondary neoplasms of subjects on both arms assessed by bone scan or axial imaging
Time Frame: From date of first dose until 30 days after the last treatment, assessed for a maximum of 24 months
Population: Data was not collected or analyzed for this objective due to the termination of the study by the funder
Arm/Group | Control Arm A | Experimental Arm B
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: PSA Complete Response Rates
Description: Subjects on both arms with PSA ≤ 0.2 ng/mL after 7 months of androgen deprivation therapy
Time Frame: From date of first dose of androgen deprivation therapy (ADT) until completion of 7 cycles (28 weeks)
Population: Data was not collected or analyzed for this objective due to the termination of the study by the funder
Arm/Group | Control Arm A | Experimental Arm B
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: PSA Partial Response Rates
Description: Subjects on both arms with PSA between 0.2 and ≤ 4 ng/mL after 7 months of androgen deprivation therapy.
Time Frame: From date of first dose of ADT until completion of 7 cycles (28 weeks)
Population: Data was not collected or analyzed for this objective due to the termination of the study by the funder
Arm/Group | Control Arm A | Experimental Arm B
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Median Time to Castration Resistance
Description: Castration resistance for subjects on both arms determined by first PSA level increase and/or radiographic progression by first imaging assessment showing progression
Time Frame: From date of ADT (first LHRH agonist/antagonist/surgical castration) to date of PSA and/or radiographic progression, assessed for a maximum of 24 months
Population: Data was not collected or analyzed for this objective due to the termination of the study by the funder
Arm/Group | Control Arm A | Experimental Arm B
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: 2-Year PSA Progression Free Survival (PFS)
Description: PSA PFS for subjects on both arms defined as first PSA level increase
Time Frame: From date of randomization to first occurrence of PSA progression, symptomatic deterioration, or death due to any cause, assessed up to 24 months
Population: Data was not collected or analyzed for this objective due to the termination of the study by the funder
Arm/Group | Control Arm A | Experimental Arm B
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: 2-Year Overall Survival (OS)
Description: OS for subjects on both arms
Time Frame: From date of randomization to death from any cause, assessed up to 24 months
Population: Data was not collected or analyzed for this objective due to the termination of the study by the funder
Arm/Group | Control Arm A | Experimental Arm B
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: 12-Week Alkaline Phosphatase (ALP) Normalization
Description: ALP normalization for subjects with abnormal ALP at randomization
Time Frame: From date of randomization until completion of 12 weeks of therapy
Population: Data was not collected or analyzed for this objective due to the termination of the study by the funder
Arm/Group | Control Arm A | Experimental Arm B
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Time to ALP Progression
Description: ALP progression of 25% or greater from baseline/nadir for subjects on both arms
Time Frame: From date of randomization until date of ALP progression, assessed up to 24 months
Population: Data was not collected or analyzed for this objective due to the termination of the study by the funder
Arm/Group | Control Arm A | Experimental Arm B
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change in Pain Over Time
Description: Subjects on both arms self-reported evaluation of worst pain item, as well as the subscale scores for pain severity and pain interference as determined by subject responses on the BPI-SF questionnaire.
Time Frame: From baseline until 30 days after the last treatment, assessed for a maximum of 24 months
Population: Data was not collected or analyzed for this objective due to the termination of the study by the funder
Arm/Group | Control Arm A | Experimental Arm B
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Analgesic Use by WHO Ladder Score
Description: Analgesic use scores for subjects on both arms will be assigned by the treating physician based on the subject's daily analgesic use on average. A single numeric score (0, 1, 2 or 3) will be assigned based on the 3-step WHO pain ladder.
Time Frame: From baseline until 30 days after the last treatment, assessed for a maximum of 24 months
Population: Data was not collected or analyzed for this objective due to the termination of the study by the funder
Arm/Group | Control Arm A | Experimental Arm B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Duration of participation in study, until study termination.
Arm/Group | Control Arm A | Experimental Arm B
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/11
Other Adverse Events (participants affected / at risk) | 4/5 | 11/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Arm A (N=5) | Experimental Arm B (N=11)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (2) | 2 (2)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (2) | 2 (2)
ANEMIA (Blood and lymphatic system disorders) | 2 (2) | 5 (8)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4)
BLOOD AND LYMPHATIC SYSTEM DISORDERS - OTHER, SPECIFY (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 3 (4) | 4 (4)
DEPRESSION (Psychiatric disorders) | 1 (1) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 1 (1) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 7 (12)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 1 (1)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (General disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 1 (2)
HOT FLASHES (Vascular disorders) | 2 (3) | 8 (8)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (1) | 4 (13)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
HYPERTENSION (Vascular disorders) | 4 (4) | 7 (12)
INSOMNIA (Psychiatric disorders) | 1 (1) | 1 (1)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 4 (5)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY (Nervous system disorders) | 1 (1) | 1 (1)
PAIN (General disorders) | 1 (1) | 3 (4)
SPASTICITY (Nervous system disorders) | 1 (1) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
URINARY URGENCY (Renal and urinary disorders) | 1 (1) | 1 (1)
AGITATION (Psychiatric disorders) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 3 (5)
AMNESIA (Nervous system disorders) | 0 (0) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ANORGASMIA (Psychiatric disorders) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 3 (4)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
CHOLESTEROL HIGH (Investigations) | 0 (0) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 0 (0) | 4 (8)
DIZZINESS (Nervous system disorders) | 0 (0) | 3 (4)
EDEMA LIMBS (General disorders) | 0 (0) | 2 (3)
EYE DISORDERS - OTHER, SPECIFY (Eye disorders) | 0 (0) | 4 (4)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
FLUSHING (Vascular disorders) | 0 (0) | 1 (1)
GYNECOMASTIA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
HEARING IMPAIRED (Ear and labyrinth disorders) | 0 (0) | 2 (2)
HEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 0 (0) | 1 (1)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS - OTHER, SPECIFY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INVESTIGATIONS - OTHER, SPECIFY (Investigations) | 0 (0) | 1 (1)
LIBIDO DECREASED (Psychiatric disorders) | 0 (0) | 1 (1)
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 (0) | 2 (2)
METABOLISM AND NUTRITION DISORDERS - OTHER, SPECIFY (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (5)
PARESTHESIA (Nervous system disorders) | 0 (0) | 1 (1)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 2 (5)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PSYCHIATRIC DISORDERS - OTHER, SPECIFY (Psychiatric disorders) | 0 (0) | 1 (1)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY (Renal and urinary disorders) | 0 (0) | 4 (4)
RENAL CALCULI (Renal and urinary disorders) | 0 (0) | 1 (1)
REPRODUCTIVE SYSTEM AND BREAST DISORDERS - OTHER, SPECIFY (Reproductive system and breast disorders) | 0 (0) | 1 (1)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SINUS BRADYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4)
SLEEP APNEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
TOOTH INFECTION (Infections and infestations) | 0 (0) | 1 (1)
URINARY FREQUENCY (Renal and urinary disorders) | 0 (0) | 5 (5)
WEIGHT GAIN (Investigations) | 0 (0) | 1 (1)
WHITE BLOOD CELL DECREASED (Investigations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated due to slow accrual. All subjects were removed from study before reaching any primary or secondary endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-09): https://cdn.clinicaltrials.gov/large-docs/49/NCT02582749/Prot_SAP_000.pdf